CLINICAL TRIAL: NCT06286852
Title: Italian Language Validation of The Eating Disorder Examination (EDE) - Child Version
Status: Active, not recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Lucilla Bonvini, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: EDE BA
Record Dates: First submitted 2024-02-15; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Feeding and Eating Disorders of Childhood
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Subjects meeting a diagnosis of nutrition and eating disorder
  Interventions: Behavioral: Administration of K-SADS-PL- Kiddie-Schedule for Affective Disorder and Schizophrenia-Present and Lifetime version (Kaufmann, 2002); Behavioral: Administration of ChEDE- Child Version of the EatingDisorder Examination
- Control group: children - adolescents from various schools in the Florence area, chosen through statistical criteria based on age, gender, ethnicity
  Interventions: Behavioral: Administration of ChEDE- Child Version of the EatingDisorder Examination

INTERVENTIONS:
Behavioral: Administration of K-SADS-PL- Kiddie-Schedule for Affective Disorder and Schizophrenia-Present and Lifetime version (Kaufmann, 2002) — Administration of 1) K-SADS-PL- Kiddie-Schedule for Affective Disorder and Schizophrenia-Present and Lifetime version (Kaufmann, 2002)
  Groups: Experimental group
Behavioral: Administration of ChEDE- Child Version of the EatingDisorder Examination — Administration of ChEDE- Child Version of the EatingDisorder Examination

SUMMARY:
Although eating disorders often occur during or after puberty, it is likely that critical antecedent conditions can be established before adolescence. The Eating Disorder Examination has been adapted for children and is described by Bryant - Waugh, Cooper, Taylor and Lask (1996). The EDE is considered the gold standard of measures of eating disorder psychopathology (Wilson, 1993), and this adaptation, which allows its use with a younger age group, is a potentially important addition to the assessment of eating disorders in children. The latest version of EDE, the l7th edition, has now surpassed its predecessors.

The aim of the study is to evaluate the psychometric properties of the Child vers ion EDE (chEDE) translated into Italian, in a sample of patients with eating disorder

ELIGIBILITY:
Inclusion Criteria:

* Subjects meet a diagnosis of nutrition and eating disorder, specifically anorexia nervosa, bulimia nervosa, binge eating disorder, according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders DSM-5
* or (for control group) Exclusion of a current or past eating disorder by performing pre-testing (KL subscales - SADS) and BMI 17.5
* Signed informed consent

Exclusion Criteria:

* Schizophrenia or other psychotic disorders;
* Substance misuse in place
* Medical complications that have the potential to hinder interpretation of results ( e.g., a medical illness that induces weight loss)
* Presence of physical treatments (including medications) that have the potential to hinder interpretation of results (e.g., chemotherapy for cancer)
* or (for control group) Presence of a current or past eating disorder and/or Ongoing eating disorder therapy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects with a diagnosis of nutrition and eating disorder, particularly anorexia nervosa, bulimia nervosa, binge eating disorder, according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders DSM-5
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
K-SADS-PL (Kiddie-Schedule for Affective Disorder and Schizophrenia-Present and Lifetime version) questionnaire | Immediately after the end of the study (last subject who will complete the qestionnaire)
  K-SADS-PL score differences between experimental group (patients with eating disorders) and control group (adolescents without eating disorders)
ChEDE (Child Version of the EatingDisorder Examination) | Immediately after the end of the study (last subject who will complete the qestionnaire)
  ChEDE score differences symptoms between patients with eating disorders and control group

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Meyer Children's Hospital IRCCS, Florence
  - USL Toscana Centro, Florence
  - Ospedale Villa Garda, Garda

IPD SHARING:
Plan to Share IPD: No